CLINICAL TRIAL: NCT03598634
Title: Epi Off Versus Epi on Corneal Collagen Cross-linking in Keratoconus Patients: a Comparative Study Throught 2 Years Follow-up
Brief Title: Epi Off Versus Epi on Corneal Collagen Cross-linking in Keratoconus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001-05-2018
Record Dates: First submitted 2018-06-12; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Keratoconus
Keywords: cross-linking
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epi-on cross-linking (Active Comparator): Intervention: Drug: Riboflavin 0.15 in 20% dextran solution
  Interventions: Procedure: administration of riboflavin for epi-off cross-linking; Procedure: administration of riboflavin for epi-on cross-linking
- Epi-off cross-linking (Active Comparator): intervention: Drug: Riboflavin 0.15 in 15% dextran solution supplemented with Tris-hydroxymethylaminomethane and sodium ethylenediaminetetraacetic acid
  Interventions: Procedure: administration of riboflavin for epi-off cross-linking; Procedure: administration of riboflavin for epi-on cross-linking

INTERVENTIONS:
Procedure: administration of riboflavin for epi-off cross-linking — riboflavin 0.1% in 20% dextran solution
Procedure: administration of riboflavin for epi-on cross-linking — riboflavin 0.1% in 15% dextran solution supplemented with tris-hydroxymethylaminomethane and sodium ethylenediminetetraacetic acid

SUMMARY:
To evaluate two different techniques of cross linking: standard epithelium off (CXL epi off) versus trans-epithelial (CXL epi on) cross linking in patient with progressive keratoconus.

DETAILED DESCRIPTION:
The aim of the study is to evaluate two different techniques of cross linking: standard epithelium off (CXL epi off) versus trans-epithelial (CXL epi on) cross linking in patient with progressive keratoconus.

Forty eyes from 32 patients with progressive keratoconus were prospectively enrolled from June 2014 to June 2015 in this non-blinded, randomized comparative study. Twenty eyes were treated by CXL epi off and 20 by CLX epi on, randomly assigned and followed for 2 years. All patients underwent a complete ophthalmologic testing that included uncorrected and best corrected visual acuity, central and peripheral corneal thickness, corneal astigmatism, simulated maximum, minimum, and average keratometry, corneal confocal microscopy, Schirmer I and break-up time (BUT) tests, and the Ocular Surface Disease Index. Intra-and postoperative complications were recorded. The solution used for CXL epi off comprised riboflavin 0.1% and dextran 20.0% (Ricrolin), whereas the solution for CXL epi on (Ricrolin, TE) comprised riboflavin 0.1%, dextran 15.0%, trometamol (Tris), and ethylene-diamine-tetra-acetic acid. Ultraviolet-A treatment was performed with UV-X System at 3 mW/cm2.

ELIGIBILITY:
Inclusion Criteria:

* patients with evolving keratoconus
* aged between 18 and 40 years
* no evidence of corneal scarring

Exclusion Criteria:

* patients with central and paracentral corneal opacities
* Vogt's striae
* previous intraocular surgery
* history of herpetic keratitis
* history of severe dry eye
* concomitant autoimmune diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity after treatment | up to 48 months from the recruitment
  * Scale name: Early treatment diabetic retinopathy study (ETDRS) charts.
  * Scale range 0-1.
  * highest value of the range (corresponding to 20/20): 0
  * lowest value of the range (corresponding to 20/200): 1

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available once the studies results will be published